CLINICAL TRIAL: NCT00801918
Title: A Phase II Pilot Multicenter Study of Denileukin Diftitox Alone and in Combination With ICE (ICED) Chemotherapy in Children, Adolescents and Young Adults (CAYA) With Relapsed or Refractory Anaplastic Large Cell Lymphoma
Brief Title: Denileukine Diftitox for Relapsed ALCL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Mitchell Cairo, MD, Prinicpal Investigator, Columbia University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC8963
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2009-10

CONDITIONS: Anaplastic Large-Cell Lymphoma
Keywords: lymphoma; pediatric; adolescent; relapsed; refractory; denileukin diftitox; Ontak
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma; Recurrence | interventions — denileukin diftitox; Ifosfamide; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DD Alone (Other): Patients will get Denileukin Diftitox for 5 days every 3 weeks for a total of 4 cycles.
  Interventions: Drug: Denileukin Diftitox
- DD with ICE Chemotherapy (Experimental): For patients who show a response to DD alone after 4 cycles or for patients who show progressive disease after 2 cycles, DD will be given with ICE chemotherapy for 2 cycles.
  Interventions: Drug: Denileukin diftitox, ifosfamide, cyclophosphamide, etoposide

INTERVENTIONS:
Drug: Denileukin Diftitox — Denileukin Diftitox: 18 mcg/kg/day: days 1-5 in cycles 1,2,3,4
  Other Names: Ontak
  Arms: DD Alone
Drug: Denileukin diftitox, ifosfamide, cyclophosphamide, etoposide — Denileukin Diftitox: 18 mcg/kg/day days 1-2 in cycles 5 and 6 Ifosfamide: 3000mg/m²/IV/d X 3 days + Mesna 3000 mg/m2/d X 3 days Carboplatin: 635mg/m2/d X 1 day Etoposide: 100mg/m2/d X 3 days
  Other Names: Ontak
  Arms: DD with ICE Chemotherapy

SUMMARY:
The purpose of this study is to determine is Denileukin diftitox will be safe, well tolerated and induce a significant overall response alone and in combination with chemotherapy: ifosfamide, carboplatin and etoposide (ICE) and will be safe and well tolerated in a population of children, adolescents and young adults with relapsed or refractory anaplastic large cell lymphoma (ALCL).

DETAILED DESCRIPTION:
Despite significant progress in the treatment and outcome for childhood ALCL, the prognosis for children who develop progressive or recurrent disease is poor with < 30% DFS. Novel therapies are urgently needed for these subgroups of patients. One potential approach is the investigation of a new class of receptor targeted cytotoxic fusion proteins (denileukin diftitox{DD}). We have previously demonstrated that > 85% of children with ALCL express CD25. The human IL-2 receptor exists in three forms, low (CD25), intermediate (CD122/CD132) and high (CD25/CD122/CD132) affinity. DD is a recombinant DNA-derived cytotoxic fusion protein composed of the amino acid sequences for diphtheria toxin fragments followed by the binding sequences for the interleukin-2 receptor. Malignant cells expressing one or more of the subunits of the IL-2 receptor are found in certain leukemias and lymphomas including cutaneous T-cell lymphoma (CTCL). Clinical studies have shown therapeutic efficacy of DD alone and in combination with CHOP chemotherapy in CD25 expressing malignancies such as CTCL, CLL and lymphoma. We hypothesize that DD will be safe and efficacious in children with relapsed ALCL.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be ≥ 2.00 year and ≤ 24.99 years of age at the time of study entry.
* Diagnosis:

Patients must have previous histologic verification of anaplastic large cell lymphoma (ALCL). Patients must be in first, second or third relapse or initial induction failure.

- Disease Status: Patients must have measurable radiographic disease.

- Performance Level: Karnofsky > 60% for patients > 16 years of age and Lansky > 60 for patients <16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

- Prior Therapy

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. Patients who are post-allogeneic transplant should be off immunosuppressive agents prior to starting therapy. Steroid doses should also be stable or decreasing for at least 1 week prior to starting therapy.

Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study (6 weeks if prior nitrosourea).

Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. These patients must be discussed with the Study Chair on a case-by-case basis.

XRT: > 2 wks for local palliative XRT (small port); > 2 months must have elapsed if prior TBI, craniospinal XRT or if > 50% radiation of pelvis; > 6 wks must have elapsed if other substantial BM radiation.

Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and > 2 months must have elapsed since SCT.

Patients may not have received prior therapy with Denileukin Diftitox

- Organ Function Requirements

Adequate Bone Marrow Function Defined As:

1. For patients without bone marrow involvement:

   * Peripheral absolute neutrophil count (ANC) > 1,000
   * Platelet count > 100,000 (transfusion independent)
   * Hemoglobin > 8.0 gm (RBC transfusion independent)
2. For patients with bone marrow involvement:

   * Peripheral absolute neutrophil count (ANC) > 1,0
   * Platelet count > 20,000 (may receive platelet transfusions)
   * Hemoglobin > 8.0 (may receive RBC transfusions)

Adequate Renal Function Defined As:

Creatinine clearance or radioisotope GFR 70mL/min/1.73m2

OR

A serum/plasma creatinine GFR calculation using the Schwartz formula (Schwartz et al. J. Peds, 106:522, 1985)

Estimated Creatinine Clearance (in mL/min/1.73 m2) = (k)(L)/Pcr

Where L = child's length in cm Pcr = plasma (or serum) creatinine (in mg/dL)

k Values = 0.33 low birth weight infant 0.45 term infant 0.55 child 0.55 adolescent female 0.70 adolescent male

Adequate Liver Function Defined As:

* Bilirubin (sum of conjugated + unconjugated) < 1.5 x upper limit of normal (ULN) for age, and
* SGPT (ALT) < 3 x upper limit of normal (ULN) for age
* Serum albumin > 2 g/dL.

Exclusion Criteria:

* Patients must not be currently receiving another investigational drug.
* Patients must not be currently receiving other anti-cancer agents.
* Patients must have a negative pregnancy test and Nursing mothers must agree not to breast-feed.
* Patients who have a documented uncontrolled infection requiring IV antibiotics
* Patients with CNS disease are not eligible.

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 5 months
Determine response rate | 6 months
Evaluate safety of combination of Denileukin Diftitox and ICE chemotherapy | 6 months

SECONDARY OUTCOMES:
Biology Studies of ALCL | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States